CLINICAL TRIAL: NCT01667224
Title: Actiponin Supplementation Reduces Abdominal Fat Area, Weight, Body Fat Mass and BMI in Obese Korean Subjects.
Brief Title: Efficacy and Safety of Actiponin on Antiobesity in Obese Korean Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TgBio-TG1022-001
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Obesity
Keywords: Actiponin; Obesity; Abdominal fat
MeSH Terms: conditions — Obesity | interventions — gypenoside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actiponin (Experimental): Actiponin(extract of Gynostema pentaphyllum, 450mg/day) for 12weeks
  Interventions: Dietary Supplement: Actiponin
- Placebo (Placebo Comparator): Placebo(450mg/day) for 12weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Actiponin — The dried leaves of G. pentaphyllum leaves were extracted with 50% ethanol and filtered; the filtrate was concentrated under high pressure and high temperature. Damulin An and B, analytical marker of Actiponin, exist more 2.49% and 1.06% respectively in raw material.
  Other Names: Extract of Gynostemma pentaphyllum(450mg/day)
  Arms: Actiponin
Dietary Supplement: Placebo — Amount and calorie of placebo are same with Actiponin.
  Other Names: Placebo(450mg/day)
  Arms: Placebo

SUMMARY:
Obesity is a major health issue worldwide; there is a constant raise in obesity related death each year. In vitro and animal studies elucidated Actiponin as a novel anti-obesity agent. However, the efficacy and safety of Actiponin supplementation on body weight regulation in humans are lacking.

DETAILED DESCRIPTION:
The primary aim of the study was to investigate the effect of Actiponin in Korean subjects on body weight and fat loss along with changes in metabolic markers based on 12 week, randomized, double-blind, placebo-controlled clinical trial.

Eighty obesity subjects with BMI > 25kg/m2 and waist-hip ratio (WHR) ≥ 0.90 for men and ≥ 0.85 for women were randomly divided into either Actiponin (n=40, 450mg/day) or placebo group (n=40, 450mg/day) for 12weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25kg/m2 and WHR ≥ 0.90(men), WHR ≥ 0.85(women)

Exclusion Criteria:

* Significant variation in weight(more 10%) in the past 3 months
* Cardiovascular disease, e.g. arrhythmia, heart failure, myocardial infarction, and patient with pacemaker
* History of disease that could interfere with the test products or impede theire absorption, such as gastrointestinal disease or gastrointestinal surgery
* Participation in any other clinical trials within past 2 months
* Abdominal hepatic liver function
* Renal disease, e.g. acute/chronic renal failure, nephritic syndrome
* Used antipsychosis drugs therapy within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnancy or breast feeding
* History of alcohol or substance abuse
* Allergic or hypersensitive to any of the ingredients in the test products

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Wan Chae, Ph.D, MD, Study Chair — Chonbuk National University Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study subjects were recruited from Clinical Trial Center for Functional Food in Chonbuk National University Hospital during the 2009. Only those subjects who were obese[both BMI≥25kg/m2 and WHR≥0.90(men), WHR≥0.85(women)] and were not diagnosed with any disease were included in this study.
Pre-assignment Details: Among the 105 subjets screened, 25 subjects had anthropometric and/or laboratory tests results that were in the exclusion criteria category, hence they were excluded from the study.
Groups:
- Actiponin: Actiponin(extract of Gynostema pentaphyllum, 450mg/day) for 12weeks
  Actiponin : The dried leaves of G. pentaphyllum leaves were extracted with 50% ethanol and filtered; the filtrate was concentrated under high pressure and high temperature. Damulin An and B, analytical marker of Actiponin, exist more 2.49% and 1.06% respectively in raw material.
- Placebo: Placebo(450mg/day) for 12weeks
  Placebo : Amount and calorie of placebo are same with Actiponin.
Period: Overall Study
Arm/Group | Actiponin | Placebo
Started | 40 | 40
Completed | 36 | 38
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Actiponin | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.10 (9.67) | 40.05 (11.58) | 40.08 (10.60)
Gender [Count of Participants; unit: Participants]
  Female | 18 | 30 | 48
  Male | 22 | 10 | 32
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Fat Mass.
Description: Body fat mass was measured in study visit 1(0 week), visit 2(4 week), visit 3(8 week) and visit 4(12 week).
Time Frame: study visit 1(0 week), visit 2(4 week), visit 3(8 week) and visit 4(12 week)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Actiponin | Placebo
Number analyzed (Participants) | 40 | 40
kg
  0 week | 22.65 (3.12) | 23.04 (3.55)
  4 week | 22.28 (3.45) | 23.17 (3.61)
  8 week | 21.89 (3.35) | 23.15 (3.8)
  12 week | 21.4 (3.62) | 23.32 (3.82)
Statistical Analysis 1: Comparison: Actiponin vs Placebo; Data are present as the mean±S.E. to detect a 0.3kg(S.D.=0.6kg) difference in body weight between groups with 80% power and a two-tailed α-value of 0.05; Test type: Non-Inferiority or Equivalence — Data are present as the mean±S.E. to detect a 0.3kg(S.D.=0.6kg) difference in body weight between groups with 80% power and a two-tailed α-value of 0.05; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Changes in Abdominal Total Fat Area.
Description: Abdominal total fat area was measured in study visit 1(0 week) and visit 4(12 week).
Time Frame: study visit 1(0 week), visit 4(12 week)
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | Actiponin | Placebo
Number analyzed (Participants) | 40 | 40
cm^2
  Pre | 332.24 (10.65) | 335.36 (7.24)
  Post | 311.35 (9.04) | 333.05 (8.36)
Statistical Analysis 1: Comparison: Actiponin vs Placebo; Data are present as the mean±S.D. to detect a 0.3kg(S.E.=0.6kg) difference in body weight between groups with 80% power and a two-tailed α-value of 0.05; Test type: Non-Inferiority or Equivalence — Data are present as the mean±S.D. to detect a 0.3kg(S.E.=0.6kg) difference in body weight between groups with 80% power and a two-tailed α-value of 0.05; p < 0.05, Mixed Models Analysis

3. Secondary Outcome: Changes in Body Weight.
Description: Body weight was measured in study visit 1(0 week), visit 2(4 week), visit 3(8 week) and visit 4(12 week).
Time Frame: study visit 1(0 week), visit 2(4 week), visit 3(8 week), and visit 4(12 week)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Actiponin | Placebo
Number analyzed (Participants) | 40 | 40
kg
  0 week | 76.56 (8.31) | 73.41 (9.79)
  4 week | 76.26 (8.35) | 73.53 (9.79)
  8 week | 75.57 (8.18) | 73.33 (9.98)
  12 week | 75.21 (8.2) | 73.33 (10.17)
Statistical Analysis 1: Comparison: Actiponin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.05, Mixed Models Analysis

4. Secondary Outcome: Changes in Body Mss Index(BMI)
Description: BMI was measured in study visit 1 (0 week), visit 2 (4 week), visit 3 (8 week) and visit 4 (12 week).
Time Frame: study visit 1(0 week), visit 2(4 week), visit 3(8 week) and visit 4(12 week)
Measure: Mean (Standard Error); unit: kg/m^2
Groups:
- Actiponin(450mg/Day) for 12week: Actiponin : The dried leaves of G. pentaphyllum leaves were extracted with 50% ethanol and filtered; the filtrate was concentrated under high pressure and high temperature. Damulin An and B, analytical marker of Actiponin, exist more 2.49% and 1.06% respectively in raw material.
- Placebo (450mg/Day) for 12 Week: Placebo: Amount and calorie of placebo are same with Actiponin
Arm/Group | Actiponin(450mg/Day) for 12week | Placebo (450mg/Day) for 12 Week
Number analyzed (Participants) | 40 | 40
kg/m^2
  0 week | 27.8 (1.21) | 27.55 (1.27)
  4 week | 27.69 (1.17) | 27.61 (1.36)
  8 week | 27.44 (1.28) | 27.54 (1.45)
  12 week | 27.31 (1.24) | 27.55 (1.54)
Statistical Analysis 1: Comparison: Actiponin(450mg/Day) for 12week vs Placebo (450mg/Day) for 12 Week; Data are present as the mean±S.E. to detect a 0.3kg(S.D.=0.60kg) difference in body weight between groups with 80% power and a two-tailed α-value of 0.05; Test type: Non-Inferiority or Equivalence — Data are present as the mean±S.E. to detect a 0.3kg(S.D.=0.60kg) difference in body weight between groups with 80% power and a two-tailed α-value of 0.05; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Actiponin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No